CLINICAL TRIAL: NCT04225169
Title: The Effect of Breathing Exercise on Pain, Anxiety, and Depression
Brief Title: The Effect of Diaphragmatic Breathing Exercise on Pain, Anxiety, and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Figen EROL URSAVAŞ, Faculty of Health Science, Department of Surgical Nursing, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CankırıKU
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Breathing Exercises
Keywords: Pain; Anxiety; Depression
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises (Experimental): diaphragmatic breathing exercises
  Interventions: Other: Breathing exercises
- Control (No Intervention): Patients in the control group received routine patient care consisting of cold therapy

INTERVENTIONS:
Other: Breathing exercises — The patient was taken to a quiet room and asked to lie on the bed. For the first 5 minutes, the researchers explained how the exercise is done with pictures and demonstrated it to the patient. The patient was asked to perform the exercise for 5 minutes under supervision by the researchers. If the patient performed DBE correctly, practice was discontinued. If not, the patient was asked to practice for another 5 minutes. If the patient still could not perform the exercise correctly at the end of this time, they were excluded from the sample. DBE was performed according to the Cleveland Clinic guideline as follows:
  Arms: Exercises

SUMMARY:
Background: After total knee replacement (TKR) surgery, patients often experience intense levels of pain, stress, and anxiety that can adversely affect postoperative recovery. Diaphragmatic breathing exercise (DBE) may help patients manage pain and emotional distress.

Aim: The aim of this study was to investigate the effect of DBE on pain, anxiety, and depression in patients undergoing TKR.

Methods: The study population consisted of patients who underwent TKR surgery in the orthopedic ward of Çankırı State Hospital between May and August 2019. The study sample included a total of 38 patients satisfying the inclusion criteria. Stratified randomization was used to assign the patients into sex-matched intervention group (n=19) and control group (n=19). Patients in the intervention group were also trained in the DBE procedure. Pain scores were evaluated at 1, 2, 4, 8, 12, and 24 hours postoperatively, while the anxiety and depression was applied on the postoperative day 2. Data were analyzed using descriptive statistics, Chi-square test, and Mann-Whitney U test.

DETAILED DESCRIPTION:
TKR is one of the most common orthopedic surgical procedures. Because TKR involves extensive muscle and bone repair, it is known to be one of the most painful operations. Moreover, as prosthetic surgery is an elective procedure, patients delay and experience anxiety about surgery due to their experiences with severe pain. This leads to chronic fear of pain and negative thought patterns. Inadequate use of analgesics and poor pain management after surgery can cause delayed mobilization, increased risk of venous thrombosis, insufficient wound healing, prolonged hospital stay, unnecessary psychological distress, and lower patient satisfaction. Many patients experience psychological problems such as depression, anxiety, discouragement, negative feelings, crying, frustration, lack of motivation, fatigue, moodiness, irritability, despair, and helplessness. Patients have expressed a need for social or psychological support. In order for patients to avoid such pain-related complications, they must be taught how to cope with pain.

The severe pain, anxiety, and stress patients experience following TKR surgery may impact their postoperative recovery. Studies have shown that nonpharmacological interventions for postoperative pain reduce pain intensity and opioid use. One of these nonpharmacological methods is diaphragmatic breathing exercises (DBE). Also known as diaphragmatic breathing or deep breathing, DBE is an effective holistic mind-body training to cope with stress and psychosomatic conditions. DBE involves contraction of the diaphragm and expansion of the belly to deepen inhalation and exhalation, which consequently decreases breathing rate and maximizes blood gas concentrations.

DBE plays an important role in pain signaling, autonomic activation, emotional regulation, acid-base equilibrium, and anti-inflammatory processes. DBE has been shown to enhance emotions, effectively reduce anxiety and its symptoms, and alleviate negative emotions such as depression, stress, and anger. There are few studies in the literature on the effect of DBE on patients who underwent TKR. One of these is a semi-experimental study that evaluated the effect of relaxation intervention (breathing exercises and guided imagery) on patients who underwent TKR. They authors reported that relaxation techniques were effective in managing patients' pain and anxiety. Another study evaluating the effect of relaxation techniques and back massage in patients who underwent TKR and total hip replacement (THR) showed that these techniques reduced patients' pain and anxiety during bedrest. Investigated the effect of a DBE program in patients with OA and found that DBE had no effect in alleviating pain or improving physical function.

A few studies have used DBE to prevent pain and sensory tension in patients who underwent TKR. However, different relaxation techniques were used in addition to DBE in these studies. To the best of our knowledge, no studies have examined the efficacy of DBE alone. Given the rising incidence of TKR, it is imperative that we strengthen our arsenal of effective interventions against the pain and psychological problems associated with this procedure. The aim of the present study was to evaluate the effect of DBE on pain, anxiety, and depression in patients who underwent TKR.

ELIGIBILITY:
Inclusion Criteria:

* Having total knee replacement

Exclusion Criteria:

* Dementia,
* Alzheimer's disease,
* Chronic obstructive pulmonary disease,
* Psychiatric disorders,
* hearing problems that prevented communication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — In light of population-based research demonstrating higher prevalence of pain among women (Fillingim et al., 2009), the patients were first stratified by sex. Block randomization was then performed by coin-flipping method to assign the patients in equal numbers to one of the two study groups.
Enrollment: 38 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Comparison of mean postoperative pain scores of patients in the intervention and control groups | The intervention and control groups completed the VAS (Visuel Analog Scale) was applied at postoperative 1, 2, 4, 8, 12, and 24 hours
  Visuel Analog Scale (VAS) This one-dimensional measure of pain intensity is a reliable and easily applicable scale that is widely accepted in the literature. VAS is used to convert nonmeasurable variables into numeric values. The 10-cm scale is labeled 0 ("no pain") at one end and 10 ("extreme pain") at the other, with values indicated at each cm in between
Comparison of mean postoperative anxiety and depression scores of patients in the intervention and control groups | HADS (Hospital Anxiety Depression Scale) was used on postoperative day 2
  Hospital Anxiety Depression Scale (HADS) The scale consists of 14 items, 7 of which assess signs of depression and 7 that assess signs of anxiety. Responses are evaluated on 4-point Likert-type scale scored between 0 and 3. However, responses to the even-numbered items decrease in severity and are scored from 3 to 0, while responses to the odd-numbered items are scored from 0 to 3. The sum of the odd-numbered items gives the anxiety score and the sum of the even-numbered items gives the depression score. The total score is not calculated. Minimum score 0, maximum score 42 higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Erol Ursavaş, Dr, Study Chair — Çankırı Karatekin University
Locations (1):
- Cankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim YC, Yobas P, Chen HC. Efficacy of relaxation intervention on pain, self-efficacy, and stress-related variables in patients following total knee replacement surgery. Pain Manag Nurs. 2014 Dec;15(4):888-96. doi: 10.1016/j.pmn.2014.02.001. Epub 2014 Jun 21. PMID 24957817
- [Background] Gatlin CG, Schulmeister L. When medication is not enough: nonpharmacologic management of pain. Clin J Oncol Nurs. 2007 Oct;11(5):699-704. doi: 10.1188/07.CJON.699-704. PMID 17962177
- [Background] Pellino TA, Gordon DB, Engelke ZK, Busse KL, Collins MA, Silver CE, Norcross NJ. Use of nonpharmacologic interventions for pain and anxiety after total hip and total knee arthroplasty. Orthop Nurs. 2005 May-Jun;24(3):182-90; quiz 191-2. doi: 10.1097/00006416-200505000-00005. PMID 15928526
- [Background] Lehrer P, Karavidas MK, Lu SE, Coyle SM, Oikawa LO, Macor M, Calvano SE, Lowry SF. Voluntarily produced increases in heart rate variability modulate autonomic effects of endotoxin induced systemic inflammation: an exploratory study. Appl Psychophysiol Biofeedback. 2010 Dec;35(4):303-15. doi: 10.1007/s10484-010-9139-5. PMID 20635134
- [Background] Busch V, Magerl W, Kern U, Haas J, Hajak G, Eichhammer P. The effect of deep and slow breathing on pain perception, autonomic activity, and mood processing--an experimental study. Pain Med. 2012 Feb;13(2):215-28. doi: 10.1111/j.1526-4637.2011.01243.x. Epub 2011 Sep 21. PMID 21939499
- [Background] Chalaye P, Goffaux P, Lafrenaye S, Marchand S. Respiratory effects on experimental heat pain and cardiac activity. Pain Med. 2009 Nov;10(8):1334-40. doi: 10.1111/j.1526-4637.2009.00681.x. Epub 2009 Aug 7. PMID 19671085
- [Background] Hayama Y, Inoue T. The effects of deep breathing on 'tension-anxiety' and fatigue in cancer patients undergoing adjuvant chemotherapy. Complement Ther Clin Pract. 2012 May;18(2):94-8. doi: 10.1016/j.ctcp.2011.10.001. Epub 2011 Nov 9. PMID 22500846
- [Background] Park E, Oh H, Kim T. The effects of relaxation breathing on procedural pain and anxiety during burn care. Burns. 2013 Sep;39(6):1101-6. doi: 10.1016/j.burns.2013.01.006. Epub 2013 Feb 1. PMID 23375536
- [Background] Larsen KL, Brilla LR, McLaughlin WL, Li Y. Effect of Deep Slow Breathing on Pain-Related Variables in Osteoarthritis. Pain Res Manag. 2019 Jun 3;2019:5487050. doi: 10.1155/2019/5487050. eCollection 2019. PMID 31281558
- [Background] Buyukyilmaz F, Asti T. The effect of relaxation techniques and back massage on pain and anxiety in Turkish total hip or knee arthroplasty patients. Pain Manag Nurs. 2013 Sep;14(3):143-54. doi: 10.1016/j.pmn.2010.11.001. Epub 2011 Jan 28. PMID 23972865